CLINICAL TRIAL: NCT02668198
Title: Diagnostic Accuracy of Using Colonoscope With Near Focus Capability in Detecting Residual Colorectal Neoplastic Tissue After Endoscopic Mucosal Resection (EMR): a Prospective Study
Brief Title: Assessing a Endoscopic Mucosal Resection Site Using Different Endoscopic Imaging Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Wallace (Other)
Collaborators: Olympus America, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Michael Wallace, Consultant, Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-007241
Record Dates: First submitted 2016-01-23; First posted 2016-01-29 (Estimated); Results first posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-09

CONDITIONS: Post-endoscopic Mucosal Resection of Colon Polyps
Keywords: Endoscopic mucosal resection, residual polyp, near focus imaging
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endoscopic scar assessment (Experimental): Using endoscope with high definition white light, high definition white light with near focus, narrow band imagining, and narrow band imaging with near focus.
  Interventions: Device: Olympus CF190 Colonoscope High definition white light; Device: Olympus CF190 Colonoscope White light with near focus; Device: Olympus CF190 Colonoscope Narrow band imaging; Device: Olympus CF190 Colonoscope Narrow band imaging with near focus; Procedure: Biopsy

INTERVENTIONS:
Device: Olympus CF190 Colonoscope High definition white light — Standard endoscopic imaging technique
Device: Olympus CF190 Colonoscope White light with near focus — Near focus mode is used to closely examine the area of prior EMR site.
Device: Olympus CF190 Colonoscope Narrow band imaging — Narrow band imaging is utilized to examine the area of prior EMR.
Device: Olympus CF190 Colonoscope Narrow band imaging with near focus — NBI with near focus to help closely examine the area of prior EMR site.
Procedure: Biopsy — Biopsy to assess any evidence of residual neoplasia via standard histopathology assessment

SUMMARY:
The purpose of this study is to compare the accuracy of using different endoscopic imaging technique (white light, white light with near focus, narrow band imaging (NBI), NBI with near focus) for detection of residual neoplastic tissue at site of prior EMR

DETAILED DESCRIPTION:
Residual neoplasia after EMR is a common. Optimal surveillance protocols are not clearly defined. There is a need for better imaging modalities to evaluate for residual disease. Suspected residual tissue can be confirmed with repeat colonoscopy or can be empirically treated. However, this can lead to either frequent colonoscopy or overtreatment. This presents more cost and financial burden to the patient. With the introduction of newer colonoscopes that have near focus/zoom capability, it is important to assess whether the near focus technology offers better accuracy for detection of residual neoplastic tissue. With better accuracy to confidently rule out residual neoplasia using newer imaging modality, additional treatment or biopsy at the previous EMR may be avoided. Furthermore, the interval for surveillance colonoscopy can be lengthened.

ELIGIBILITY:
Inclusion Criteria:

* Post-EMR follow up at 6-12 months

Exclusion Criteria:

* Non-corrected coagulopathy
* Pregnancy
* Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kandel P, Brand EC, Pelt J, Ball CT, Chen WC, Bouras EP, Gomez V, Raimondo M, Woodward TA, Wallace MB; EMR SCAR Group. Endoscopic scar assessment after colorectal endoscopic mucosal resection scars: when is biopsy necessary (EMR Scar Assessment Project for Endoscope (ESCAPE) trial). Gut. 2019 Sep;68(9):1633-1641. doi: 10.1136/gutjnl-2018-316574. Epub 2019 Jan 11. PMID 30635409
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Endoscopic Scar Assessment: Using endoscope with high definition white light, high definition white light with near focus, narrow band imaging, and narrow band imaging with near focus.
  Olympus CF190 Colonoscope High definition white light: Standard endoscopic imaging technique
  Olympus CF190 Colonoscope White light with near focus: Near focus mode is used to closely examine the area of prior endoscopic mucosal resection (EMR) site.
  Olympus CF190 Colonoscope Narrow band imaging: Narrow band imaging is utilized to examine the area of prior EMR.
  Olympus CF190 Colonoscope Narrow band imaging (NBI) with near focus: NBI with near focus to help closely examine the area of prior EMR site.
  Biopsy: Endoscopic colorectal mucosal resection
Period: Overall Study
Arm/Group | Endoscopic Scar Assessment
Started | 230
Completed | 230
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Endoscopic Scar Assessment: Using endoscope with high definition white light, high definition white light with near focus, narrow band imaging, and narrow band imaging with near focus.
  Olympus CF190 Colonoscope High definition white light: Standard endoscopic imaging technique
  Olympus CF190 Colonoscope White light with near focus: Near focus mode is used to closely examine the area of prior EMR site.
  Olympus CF190 Colonoscope Narrow band imaging: Narrow band imaging is utilized to examine the area of prior EMR.
  Olympus CF190 Colonoscope Narrow band imaging with near focus: NBI with near focus to help closely examine the area of prior EMR site.
  Biopsy: Endoscopic colorectal mucosal resection
Arm/Group | Endoscopic Scar Assessment
Number analyzed (Participants) | 230
Age, Continuous [Median (Full Range); unit: years] | 65.5 [38 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 117
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 230

OUTCOME MEASURES:

1. Primary Outcome: Positive Recurrent Adenomas Using White Light Imaging
Description: The number of positive diagnoses using white light optical imaging only.
Time Frame: approximately 6 to 12 months post endoscopic mucosal resection
Measure: Number; unit: adenomas with positive diagnoses
Groups:
- Endoscopic Scar Assessment: Using endoscope with high definition white light, high definition white light with near focus, narrow band imaging, and narrow band imaging with near focus.
  Olympus CF190 Colonoscope High definition white light: Standard endoscopic imaging technique
  Olympus CF190 Colonoscope White light with near focus: Near focus mode is used to closely examine the area of prior EMR site.
  Olympus CF190 Colonoscope Narrow band imaging: Narrow band imaging is utilized to examine the area of prior EMR.
  Olympus CF190 Colonoscope Narrow band imaging with near focus: NBI with near focus to help closely examine the area of prior EMR site.
  Biopsy: Biopsy to assess any evidence of residual neoplasia via standard histopathology assessment
Arm/Group | Endoscopic Scar Assessment
Number analyzed (Participants) | 230
adenomas with positive diagnoses | 66

2. Primary Outcome: Positive Recurrent Adenomas Using White Light Imaging Confirmed by Histology
Description: The number of recurrent adenomas diagnosed positive with white light imaging confirmed by standard histopathology of biopsy.
Time Frame: approximately 6 to 12 months post endoscopic mucosal resection
Measure: Number; unit: adenomas confirmed positive diagnoses
Arm/Group | Endoscopic Scar Assessment
Number analyzed (Participants) | 230
adenomas confirmed positive diagnoses | 56

3. Primary Outcome: Positive Recurrent Adenomas Using White Light Near Focus Imaging
Description: The number of positive diagnoses using white light near focus optical imaging only.
Time Frame: approximately 6 to 12 months post endoscopic mucosal resection
Measure: Number; unit: adenomas with positive diagnoses
Arm/Group | Endoscopic Scar Assessment
Number analyzed (Participants) | 230
adenomas with positive diagnoses | 70

4. Primary Outcome: Positive Recurrent Adenomas Using White Light Near Focus Imaging Confirmed by Histology
Description: The number of recurrent adenomas diagnosed positive with white light imaging near focus confirmed by standard histopathology of biopsy.
Time Frame: approximately 6 to 12 months post endoscopic mucosal resection
Measure: Number; unit: adenomas confirmed positive diagnoses
Arm/Group | Endoscopic Scar Assessment
Number analyzed (Participants) | 230
adenomas confirmed positive diagnoses | 57

5. Primary Outcome: Positive Recurrent Adenomas Using Narrow Band Imaging
Description: The number of positive diagnoses using narrow band optical imaging only.
Time Frame: approximately 6 to 12 months post endoscopic mucosal resection
Measure: Number; unit: adenomas with positive diagnoses
Arm/Group | Endoscopic Scar Assessment
Number analyzed (Participants) | 230
adenomas with positive diagnoses | 68

6. Primary Outcome: Positive Recurrent Adenomas Using Narrow Band Imaging Confirmed by Histology
Description: The number of recurrent adenomas diagnosed positive with narrow band imaging confirmed by standard histopathology of biopsy.
Time Frame: approximately 6 to 12 months post endoscopic mucosal resection
Measure: Number; unit: adenomas confirmed positive diagnoses
Arm/Group | Endoscopic Scar Assessment
Number analyzed (Participants) | 230
adenomas confirmed positive diagnoses | 57

7. Primary Outcome: Positive Recurrent Adenomas Using Narrow Band Imaging Near Focus
Description: The number of positive diagnoses using narrow band optical imaging near focus only.
Time Frame: approximately 6 to 12 months post endoscopic mucosal resection
Measure: Number; unit: adenomas with positive diagnoses
Arm/Group | Endoscopic Scar Assessment
Number analyzed (Participants) | 230
adenomas with positive diagnoses | 70

8. Primary Outcome: Positive Recurrent Adenomas Using Narrow Band Imaging Near Focus Confirmed by Histology
Description: The number of recurrent adenomas diagnosed positive with narrow band imaging near focus confirmed by standard histopathology of biopsy.
Time Frame: approximately 6 to 12 months post endoscopic mucosal resection
Measure: Number; unit: adenomas confirmed positive diagnoses
Arm/Group | Endoscopic Scar Assessment
Number analyzed (Participants) | 230
adenomas confirmed positive diagnoses | 58

9. Primary Outcome: Positive Recurrent Adenomas Using Biopsy
Description: The number of positive diagnoses determined by standard histopathology assessment of biopsy.
Time Frame: approximately 6 to 12 months post endoscopic mucosal resection
Measure: Number; unit: adenomas with positive diagnoses
Arm/Group | Endoscopic Scar Assessment
Number analyzed (Participants) | 230
adenomas with positive diagnoses | 62

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the colonoscopy procedure, an average of 30-45 minutes over approximately 2 years.
Arm/Group | Endoscopic Scar Assessment
All-Cause Mortality (participants affected / at risk) | 0/230
Serious Adverse Events (participants affected / at risk) | 0/230
Other Adverse Events (participants affected / at risk) | 0/230

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT02668198/Prot_SAP_000.pdf